CLINICAL TRIAL: NCT03641391
Title: Prospective Study of Awake Intraoperative Language Mapping and Construction of Chinese Probabilistic Map Based on Direct Electrical Stimulation
Brief Title: Awake Intraoperative Language Mapping and Chinese Probabilistic Map Construction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Huashan Hospital North, Fudan University (Unknown)
Responsible Party: Principal Investigator, Jinsong Wu, Professor, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KY2012-009
Record Dates: First submitted 2018-08-14; First posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Glioma
Keywords: Awake surgery; Direct cortical stimulation; Language mapping; Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Direct electrical stimulation (Experimental): Intraoperative direct cortical electrical stimulation or intraoperative direct subcortical electrical stimulation on language or language-associate areas, and the participants' after-discharge activity would be monitored. The participants would be undergone awake anesthesia and asked to perform language tasks during the stimulation.
  Interventions: Procedure: Intraoperative direct cortical electrical stimulation; Procedure: Intraoperative direct subcortical electrical stimulation

INTERVENTIONS:
Procedure: Intraoperative direct cortical electrical stimulation — Intraoperative direct electrical stimulation on language or language-associate cortex, was performed using a 5-mm wide bipolar electrode with a pulse frequency of 60 Hz and an amplitude of 1.5 to 6 milliamperage. The somatosensory evoked potential was recorded with a 6-contact subdural strip electrode. If after-discharge activity indicated that the stimulation current was too high, the current amplitude was decreased by 0.5 to 1 milliamperage. The participants would be undergone awake anesthesia and asked to perform language tasks during the stimulation.
Procedure: Intraoperative direct subcortical electrical stimulation — Intraoperative direct electrical stimulation on language or language-associate subcortical pathways, was performed using a biphasic square-wave pulse delivered at 60 Hz with a current amplitude ranging from 1.5 to 10 milliamperage. The somatosensory evoked potential was recorded with a 6-contact subdural strip electrode. If after-discharge activity indicated that the stimulation current was too high, the current amplitude was decreased by 0.5 to 1 milliamperage. The participants would be undergone awake anesthesia and asked to perform language tasks during the stimulation.

SUMMARY:
The study aims at constructing a Chinese language probabilistic map by awake intraoperative direct electrical stimulation (DES) language mapping. At the same time, the standardization and optimization of awake intraoperative DES parameters will be explored, factors affecting postoperative function morbidity and survival will also be analyzed.

DETAILED DESCRIPTION:
The study aims at constructing a Chinese language probabilistic map by awake intraoperative direct electrical stimulation (DES) language mapping.

The "maximal safe resection" of brain tumor adjacent to language cortex requires precise real-time localization of the intraoperative language cortex.

Awake craniotomy combined with DES to localize language cortex has been carried out for several decades. However, there is yet no unified standard on the specification of its technical parameters. Besides, language probabilistic maps based on DES have been reported by several teams around the world. However these studies were based on the Indo-European language speakers alone. There was one paper published in 2015 by the investigators' group using DES for the Chinese probabilistic map, but it is also a single center study, and the sample size is relatively small.

Awake craniotomy and intraoperative DES for language cortex localization will be used to construct a Chinese probabilistic map in this study. Several common tasks for language mapping (i.e., number counting, picture naming, word reading) will be applied in Chinese speakers. The positive language sites including speech arrest, anomia, alexia, anarthria, dysarthria, semantic paraphasia and phonological paraphasia, spatial negativity and other higher order cognitive function will be identified in individual patients and normalized to the standard brain atlas. The corresponding probabilistic maps will be integrated and generated.

At the same time, the standardization and optimization of awake intraoperative DES parameters will be explored, factors affecting postoperative function morbidity and survival will also be analyzed.

Through this study, the investigators will further popularize individualized awake surgery of glioma in language cortex, improve the extent of tumor resection, protect postoperative language function and improve postoperative quality of life. By constructing this standardized Chinese probabilistic map, the investigators will provide more direct evidence for brain language research.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 14-70 years with highly suspected (as assessed by study surgeon), newly diagnosed, untreated malignant glioma;
2. Individuals with gliomas with bodies involving in dominate side language area(see appendix 1);
3. Individuals with the preoperative assessment that radiological radically should be achieved;
4. Individuals who are cooperative and well tolerated with awake craniotomy;
5. Individuals presents with good communicate and explanation preoperatively;
6. All participants gave written informed consent.

Appendix 1. Tumor location in eloquent areas: located in or close to areas of the dominant-hemisphere that associated with motor or language functions, including:

1. Frontal lobe, which divided into inferior frontal gyrus (BA44-Pars opercularis, BA45-Pars triangularis/Broca's area), middle frontal gyrus (BA9, BA46), superior frontal gyrus (BA4, BA6, BA8), primary motor cortex (BA4), premotor cortex (BA6), and supplementary motor area (BA6);
2. Parietal lobe, which divided into inferior parietal lobule (BA40- supramarginal gyrus, BA39-angular gyrus), parietal operculum (BA43), and primary somatosensory cortex (BA1, BA2, BA3);
3. Temporal lobe, which divided into transverse temporal gyrus (BA41, BA42), superior temporal gyrus (BA38, BA22/Wernicke's area), middle temporal gyrus (BA21);
4. Insular lobe.

Exclusion Criteria:

1. Individuals with age < 14 years or > 70 years;
2. Individuals presents with impaired cognitive function or unstable mental status;
3. Individuals has higher intracranial pressure, sleep apnea syndrome, difficult airway or morbid obesity, claustrophobia, uncontrolled coughing, uncontrolled seizures or inability to stay still etc.;
4. Recurrent gliomas after surgery (except needle biopsy);
5. Primary gliomas with history of radiotherapy or chemotherapy;
6. Renal insufficiency or hepatic insufficiency;
7. History of malignant tumors at any body site;
8. Tumors of the midline, basal ganglia, cerebellum, or brain stem;
9. Inability or unwilling to give informed consent.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of postoperative language deficits | The first month and the third month after surgery
  Language deficits were considered when the participant presents with aphasia or severe dysphasia measured by standardized Aphasia Battery of Chinese (ABC, a Chinese version of Western Aphasia Battery) having the Aphasia Quotient (AQ) less than 50 (where lower values represent a worse outcome).

SECONDARY OUTCOMES:
Location of positive sites in cortical mapping | During surgery
  Positive stimulation of the language area was assumed when the participant exhibited counting interruption, errors during object naming, language confusion or other language problems induced by DES.
  Positive stimulation of the motion area was assumed when movements of the contralateral limb, face, lip or tongue were induced by DES, with the concurrent recording of an electromyogram.
  Positive stimulation affecting the sensation area was assumed when an abnormal feeling was induced by DES in the contralateral limb, face, lip or tongue.
  The locations of positive sites will be recorded by neuro-navigation system.
Incidence rate of intraoperative epilepsy induced by direct cortical stimulation | During surgery
  A strip electrode would be placed tangentially over the central sulcus to monitor cortical seizure activity or after-discharge during intraoperative DCS. And the participant would be closely observed for involuntarily shaking or twitching. Any shaking, twitching or after-discharge during monitor would considered as epileptic event. All epileptic events will be recorded and DES will be terminated for the participant.
Extent of resection | Within 72h after surgery
  Extent of resection (EOR) based on early postoperative MRI obtained within 72h after surgery. Gross total resection (GTR) was defined as the complete disappearance of all enhancing lesions (T1WI) for HGG and the complete disappearance of all nonenhancing (T2WI FLAIR) lesions for LGG. The EOR were quantitatively volumetric analyses for all gliomas and gliomas grouped according to eloquent areas and non-eloquent areas, and stratified as: GTR, 100% resection; subtotal resection ≥ 90% resection, partial resection ≥ 70% resection, biopsy, resection ≥98% for overall survival advantage (HGG) and resection ≥90% for overall survival advantage (LGG).

CONTACTS AND LOCATIONS:
Overall Officials: Jinsong Wu, MD, Principal Investigator — Huashan Hospital; Dongxiao Zhuang, MD, Study Director — Huashan Hospital; Tianming Qiu, MD, Study Director — Huashan Hospital; Junfeng Lu, MD, Study Director — Huashan Hospital
Locations (3):
- China (3):
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Huashan Hospital North, Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided
Please refer to the principle investigator for participants' data.

REFERENCES:
- [Background] Tate MC, Herbet G, Moritz-Gasser S, Tate JE, Duffau H. Probabilistic map of critical functional regions of the human cerebral cortex: Broca's area revisited. Brain. 2014 Oct;137(Pt 10):2773-82. doi: 10.1093/brain/awu168. Epub 2014 Jun 25. PMID 24970097
- [Background] Sanai N, Mirzadeh Z, Berger MS. Functional outcome after language mapping for glioma resection. N Engl J Med. 2008 Jan 3;358(1):18-27. doi: 10.1056/NEJMoa067819. PMID 18172171
- [Background] Chang EF, Breshears JD, Raygor KP, Lau D, Molinaro AM, Berger MS. Stereotactic probability and variability of speech arrest and anomia sites during stimulation mapping of the language dominant hemisphere. J Neurosurg. 2017 Jan;126(1):114-121. doi: 10.3171/2015.10.JNS151087. Epub 2016 Feb 19. PMID 26894457
- [Background] Duffau H. Stimulation mapping of white matter tracts to study brain functional connectivity. Nat Rev Neurol. 2015 May;11(5):255-65. doi: 10.1038/nrneurol.2015.51. Epub 2015 Apr 7. PMID 25848923
- [Background] Wu J, Lu J, Zhang H, Zhang J, Yao C, Zhuang D, Qiu T, Guo Q, Hu X, Mao Y, Zhou L. Direct evidence from intraoperative electrocortical stimulation indicates shared and distinct speech production center between Chinese and English languages. Hum Brain Mapp. 2015 Dec;36(12):4972-85. doi: 10.1002/hbm.22991. Epub 2015 Sep 9. PMID 26351094
- [Background] Wu J, Lu J, Zhang H, Zhang J, Mao Y, Zhou L. Probabilistic map of language regions: challenge and implication. Brain. 2015 Mar;138(Pt 3):e337. doi: 10.1093/brain/awu247. Epub 2014 Sep 4. No abstract available. PMID 25190682
- [Background] Nakai Y, Jeong JW, Brown EC, Rothermel R, Kojima K, Kambara T, Shah A, Mittal S, Sood S, Asano E. Three- and four-dimensional mapping of speech and language in patients with epilepsy. Brain. 2017 May 1;140(5):1351-1370. doi: 10.1093/brain/awx051. PMID 28334963
- [Background] Breshears JD, Molinaro AM, Chang EF. A probabilistic map of the human ventral sensorimotor cortex using electrical stimulation. J Neurosurg. 2015 Aug;123(2):340-9. doi: 10.3171/2014.11.JNS14889. Epub 2015 May 15. PMID 25978714
- [Background] Lu J, Wu J, Yao C, Zhuang D, Qiu T, Hu X, Zhang J, Gong X, Liang W, Mao Y, Zhou L. Awake language mapping and 3-Tesla intraoperative MRI-guided volumetric resection for gliomas in language areas. J Clin Neurosci. 2013 Sep;20(9):1280-7. doi: 10.1016/j.jocn.2012.10.042. Epub 2013 Jul 10. PMID 23850046
- [Background] Ritaccio AL, Brunner P, Schalk G. Electrical Stimulation Mapping of the Brain: Basic Principles and Emerging Alternatives. J Clin Neurophysiol. 2018 Mar;35(2):86-97. doi: 10.1097/WNP.0000000000000440. PMID 29499015